CLINICAL TRIAL: NCT05898828
Title: Phase I/II Evaluation of a Cancer Lysate Vaccine and Montanide(R) ISA-51 VG With Entinostat and Nivolumab as Adjuvant Therapy Following Chemoradiation Therapy With or Without Surgery for Locally Advanced Esophageal Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No enrollment
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001544; 001544-C
Record Dates: First submitted 2023-06-09; First posted 2023-06-12 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Neoplasms; Esophageal Neoplasms; Esophagus Neoplasm; Esophagus Cancer; Neoplasms, Esophageal; Esophageal Cancer (EsC)
Keywords: Cell Mediated Response; immune subsets; peripheral immune subsets; CT antigens; neoadjuvant chemoradiation therapy (nCRT); H1299 Cell Lysates; EsC; Immunotherapy
MeSH Terms: conditions — Neoplasms; Esophageal Neoplasms | interventions — Nivolumab; entinostat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ Phase I (Experimental): H1299 cell lysate vaccine with Montanide(R) ISA-51 VG, entinostat, and nivolumab (Phase I component to determine lysate dose)
  Interventions: Drug: Nivolumab; Drug: Entinostat; Biological: Montanide(R) ISA-51 VG Adjuvant; Biological: H1299 Cell Lysates
- 2/ Phase II (Experimental): H1299 cell lysate vaccine with Montanide(R) ISA-51 VG, entinostat, and nivolumab (lysate at dose determined in Phase I)
  Interventions: Drug: Nivolumab; Drug: Entinostat; Biological: Montanide(R) ISA-51 VG Adjuvant; Biological: H1299 Cell Lysates

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 480 mg flat dose via intravenous infusion on Day 3 of every cycle starting at Cycle 2, for intended duration of 1 year.
Drug: Entinostat — Entinostat (5 mg) self-administered on Days -14 and -7 prior to the first vaccination cycle, then entinostat (3 mg) self-administered on Days 1, 8, 15, and 22 of each vaccine cycle (Cycles 1-6). Entinostat continuation for subjects with immunologic response and NED during additional 2 vaccine injections.
Biological: Montanide(R) ISA-51 VG Adjuvant — H1299 cell lysate with Montanide(R) ISA-51 VG adjuvant vaccine via subcutaneous injections once every cycle (1 cycle=28 days) for 6 cycles (i.e., 6 vaccinations). Dose Level 1 (DL1) starting dose is 20 mg lysate protein in 2-2.5 mL Montanide(R) ISA-51 VG adjuvant; lysate concentration will be 8-10 mg/mL. Additional 2 vaccine injections for subjects with immunologic response and NED.
Biological: H1299 Cell Lysates — H1299 cell lysate with Montanide(R) ISA-51 VG adjuvant vaccine via subcutaneous injections once every cycle (1 cycle=28 days) for 6 cycles (i.e., 6 vaccinations). Dose Level 1 (DL1) starting dose is 20 mg lysate protein in 2-2.5 mL Montanide(R) ISA-51 VG adjuvant; lysate concentration will be 8-10 mg/mL. Additional 2 vaccine injections for subjects with immunologic response and NED.

SUMMARY:
This is a Phase I/II study to determine the safety and immune response of the H1299 cell lysate vaccine mixed with Montanide(R) ISA-51 VG adjuvant, to be administered on the study in combination with Entinostat and Nivolumab in eligible participants with locally advanced esophageal cancers (EsC) following either neoadjuvant chemoradiation therapy (nCRT) or nCRT and surgery. Phase I of the protocol aims to determine the safe dose of the H1299 lung cancer cell lysate vaccine mixed with Montanide(R) ISA-51 VG adjuvant when it is administered in combination with Entinostat and Nivolumab. Phase II of the protocol will focus on assessing the level of immune response in participants receiving the study intervention when the H1299 cell lysate vaccine with Montanide(R) ISA-51 VG adjuvant is administered at the dose level determined in Phase I.

DETAILED DESCRIPTION:
Background:

* Esophageal cancers (EsC) are highly lethal malignancies with strong predilections for local and systemic recurrences despite aggressive multimodality interventions.
* Currently the standard of care for locally advanced (stage II/III) EsC is neoadjuvant chemoradiation therapy (nCRT) and surgery.
* Nearly 50% of patients with esophageal squamous cell cancers (ESCC) and 25% of patients with esophageal adenocarcinomas (EAC) have pathologic complete responses (pCR) following nCRT.
* Current staging modalities cannot reliably detect all residual EsC following nCRT, and the benefit of surgery in patients with pCR is unclear.
* Recently nivolumab was approved as adjuvant therapy for patients who have undergone complete (R0) resections of locally advanced esophageal or gastro-esophageal junction (GEJ) carcinomas with pathologic incomplete responses (pIR) following nCRT.
* Preclinical studies and early phase clinical studies suggest that immune checkpoint inhibitors can improve the efficacy of vaccines targeting tumor associated antigens.
* Cancer-testis (CT) antigens (CTA), particularly those encoded by genes on the X chromosome (CT-X antigens) have emerged as attractive targets for cancer immunotherapy given their highly restricted expression in cancers but not normal tissues and oncogenic activities.
* Recent studies suggest that CT antigens are preferentially expressed in pluripotent stem/tumor initiating cells that mediate treatment resistance and metastasis of human cancers.
* Treatment interventions that inhibit activity of immunosuppressive Treg cells significantly increase efficacy of cancer vaccines and immune checkpoint inhibitors; the triple combination therapy cures nearly all mice with established, highly aggressive cancers.
* The class I histone deacetylase (HDAC) inhibitor, entinostat which inhibits Treg activity appears to favorably modulate immune cell subsets in patients with advanced cancers receiving nivolumab.
* Conceivably, vaccination of EsC patients with tumor cell lysates containing high levels of CT antigens in combination with entinostat will facilitate eradication of dormant EsC cells following immune checkpoint blockade.

Primary Objectives:

* Phase I: To determine the safe dose of adjuvant H1299 lung cancer cell lysate vaccines with Montanide(R) ISA-51 VG administered in conjunction with entinostat and nivolumab in participants with locally advanced esophageal cancers (EsC) with pathologic incomplete responses (pIR) following neoadjuvant chemoradiation therapy (nCRT).
* Phase II: To assess the frequency of immunologic responses to purified CT antigens in EsC participants following vaccinations with H1299 cancer cell lysates and Montanide(R) ISA- 51 VG in combination with entinostat and nivolumab.

Eligibility:

* Participants with clinical Stage II or Stage III EsC with pIR following nCRT within the past 16 weeks
* Participants must be 18 years or older with an ECOG performance status of 0 1
* Adequate bone marrow, kidney, liver, lung, and cardiac function
* No prior anti-PD-1/PD-L1 therapy for their EsC
* Participants receiving steroids at supraphysiologic doses will be excluded.
* Participants with HIV or any active infections will be excluded.

Design:

* After recovery from nCRT or nCRT and surgery, eligible participants will commence oral entinostat (5 mg q week).
* Following a two-week entinostat run-in, participants will commence monthly deep subcutaneous vaccinations with H1299 cell lysates and Montanide (r) ISA-51 VG until six vaccinations have been given (each cycle=28 days).
* Following the two-week entinostat (5 mg q week) run-in, entinostat will be administered at a dose of 3 mg q week during nivolumab therapy.
* Four weeks after the first vaccination, participants will commence nivolumab (480 mg IV infusion) monthly for 1 year.
* Each cycle of vaccine therapy is 4 weeks (28 days).
* Participants will be scanned every 12 weeks while on treatment or continued treatment, and during follow up every 3 months for 3 years, every 6 months for another 2 years or through disease progression.
* Leukapheresis will be performed at baseline and at treatment evaluation one month following completion of the six vaccinations.
* Systemic toxicities and immunologic responses to therapy will be recorded.
* Pre- and post-vaccination serologic and cell mediated responses to a panel of CT antigens will be assessed before and one month following completion of the six vaccinations.
* Individuals deemed to have responded to the vaccine regimen and exhibit no evidence of disease recurrence or secondary malignancy will be eligible for two additional vaccinations administered q3 months with weekly entinostat and monthly nivolumab.
* Numbers and percentages of immune subsets, soluble factors, and cytokines in peripheral blood will be assessed before and after the six vaccinations.
* Immunologic responses to autologous tumor cells (if available) as well as lysates from H1299 cells and EsC stem cells vs normal esophageal-induced pluripotent stem cells (Eso-iPSC) will be evaluated in an exploratory manner.
* Accrual ceiling will be set at 50 participants.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants with clinical Stage II (T2/N0-N1; T3/N0) or Stage III (T1-T2/N2, T3/N1-N2) EsC per 8th edition TNM Staging System who have histologically documented or suspected residual disease in the esophagus or regional nodes following nCRT. Diagnosis must be confirmed by the NIH Laboratory of Pathology.
* No prior anti-PD1/anti-PD-L1 therapy for their EsC.
* Participant must be enrolled within 16 weeks following completion of nCRT or nCRT/surgery
* ECOG performance status of 0-1.
* 18 years of age or older
* Participant must be willing to co-enroll on 06C0014 (Prospective Analysis of Genetic and Epigenetic Alterations in Patients with Thoracic Malignancies) allowing for the use of tumor or normal tissues for correlative experiments pertaining to this protocol and related translational research efforts in the Thoracic Surgery Branch (TSB).
* Adequate bone marrow reserve, hepatic and renal function as evidenced by the following laboratory parameters (all eligibility assessment/enrollment bloodwork must be done at NIH no more than 2 weeks prior to initiation of study therapy):

  * Absolute neutrophil count greater than 1500/mm^3
  * Platelet count greater than 100,000/mm^3
  * Hemoglobin greater than 8 g/dL (participants may receive transfusions to meet this parameter)
  * INR <= 1.5 x ULN
  * Total bilirubin <1.5 x upper limits of normal (except those with Gilberts disease)
  * Serum creatinine less than or equal to 1.6 mg/mL or the eGFR (calculated per institutional standards) must be greater than 60 mL/min/1.73m^2
* Oxygen saturation equal to or greater than 92% on room air within 2 weeks of initiation of study therapy.
* Seronegative for HIV antibody by bloodwork performed at NIH no more than 4 weeks prior to initiation of study therapy.
* Seronegative for active hepatitis B, and seronegative for hepatitis C antibody by bloodwork performed at NIH no more than 4 weeks prior to initiation of study therapy. If hepatitis C antibody test is positive, then participant must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) within 28 days prior to initiation of study therapy, for the duration of study participation and up to 5 months after the last dose of study therapy.
* Participants who are breastfeeding or plan to breastfeed must agree to discontinue/postpone breastfeeding while receiving investigational treatment and for 5 months after the last dose study therapy.
* Participants must be able to understand and willing to sign an informed consent.

EXCLUSION CRITERIA:

* Participants who are receiving any other investigational agents
* Participants with a history of pneumonitis will be excluded unless cleared by Pulmonary Medicine consultants
* Participants requiring chronic systemic treatment with steroids above physiologic doses.
* Participants receiving warfarin anticoagulation, who cannot be transitioned to other agents such as enoxaparin or dabigatran, and for whom anticoagulants cannot be held for up to 24 hours.
* Participants with uncontrolled hypertension (>160/95) at screening, unstable coronary disease evidenced by EKG evidence of cardiac ischemia or uncontrolled arrhythmias, unstable angina, decompensated CHF (>NYHA Class II), or myocardial infarction within 6 months prior to initiation of study therapy.
* Participants with any of the following pulmonary function abnormalities: FEV, < 35% predicted; DLCO < 35% predicted (post-bronchodilator); based on assessment performed no more than 4 weeks prior to initiation of study therapy.
* Participant pregnancy.
* Other malignancy requiring treatment with the exception of localized skin cancer amenable to topical therapies
* Uncontrolled intercurrent illness occurring within 3 months prior to initiation of study therapy that would limit compliance with study requirements. Intercurrent illness may include any conditions uncovered during screening assessments (physical examination, laboratory assessments, etc.) that, in the judgment of the investigator, precludes participation because it could present disproportionate risk to the participant

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Phase I Component: To determine the safe dose of adjuvant H1299 lung cancer cell lysate vaccines with Montanide(R) ISA-51 VG administered in conjunction with entinostat and nivolumab in participants with locally advanced esophageal cancers (EsC)... | before each cycle, every 2 weeks during Cycles 1 and 2 (AE only), at each treatment evaluation, and at the safety visit
  Assessment of safety and tolerability as determined by the frequency and severity of adverse events
Phase II Component: To assess the frequency of immunologic responses to purified cancer-testis (CT) antigens in EsC participants receiving adjuvant vaccinations with H1299 cell lysate/Montanide(R) ISA-51 VG in combination with entinostat and niv... | within 2 weeks prior to initiation of treatment, prior to 1st vaccination, 1 month following first 6 vaccinations, and every 6 months (24 weeks) during treatment continuation
  Assessment of immune response to CT antigens (new serologic reactivity or increase in existing antibody response to CT antigens, evidenced by IgM/IgG class switch or antibody titer)

SECONDARY OUTCOMES:
Phase I Component: To assess the frequency of immunologic responses to purified cancer-testis (CT) antigens in EsC participants receiving adjuvant vaccinations with H1299 cell lysate/Montanide(R) ISA-51 VG in combination with entinostat and nivo... | within 2 weeks prior to initiation of treatment, prior to 1st vaccine, one month following the first six vaccinations (start of cycle 7), and every 6 months (24 weeks) during treatment continuation
  Analyses which investigate immunologic response (i.e., immune response to CT antigens); response to vaccine will be the appearance of new serologic reactivity or an increase in existing antibody response to CT antigens, evidenced by IgM/IgG class switch or antibody titer.
Phase I + II Component: To assess safety of adjuvant H1299 lung cancer cell lysate vaccines with Montanide(R) ISA-51 VG administered in conjunction with entinostat and nivolumab in participants with locally advanced esophageal cancers (EsC) with... | before each cycle, every 2 weeks between vaccines 1 and 2, at each treatment evaluation, and at the safety visit
  Assessment of safety and tolerability as determined by the frequency and severity of adverse events
Phase II Component: To determine progression free survival (PFS) in EsC participants receiving the investigational adjuvant vaccine regimen | every 12 weeks while on treatment or continued treatment, and during follow up every 3 months for 3 years, every 6 months for another 2 years or through disease progression ending at time of final PFS evaluation at 5 years post-enrollment
  Progression free survival (PFS) determined by RECIST using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded will be shared upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers after the trial has been completed and closed.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001544-C.html